CLINICAL TRIAL: NCT04326829
Title: A Single-arm, Multi-center, Phase Ⅱ Clinical Study to Evaluate Efficacy and Safety of QL1604 Monotherapy for the Treatment of Unresectable or Metastatic Mismatch Repair Deficient (dMMR) or Microsatellite Instability-high (MSI-H) Solid Tumors That Failed to Respond to Standard Therapy
Brief Title: QL1604 Monotherapy for dMMR or MSI-H Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1604-201
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1604 Injection (Experimental)
  Interventions: Drug: QL1604

INTERVENTIONS:
Drug: QL1604 — QL1604, IV infusion

SUMMARY:
In this study, patients with previously-treated locally-advanced or metastatic mismatched repair deficient (dMMR) or microsatellite instability-high (MSI-H) colorectal carcinoma (CRC) and other solid tumors will be treated with QL1604 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF);
2. Age ≥ 18 years and ≤ 80 years when ICF is signed;
3. Histologically confirmed locally advanced or metastatic dMMR or MSI-H status colorectal carcinoma or other malignant solid tumors;
4. At least one measureable lesion as defined per RECIST Version (v) 1.1 ;
5. Subjects who have disease progression or intolerable reactions after the currently available standard anti-cancer treatment previously received or refused prior cancer therapy regimen(s) ;
6. Subjects must provide tumor tissues and blood samples for the determination of MSI, tumor mutational burden (TMB), PD-L1 expression level;
7. Eastern Cooperative Oncology Group performance status of 0 or 1;
8. Life expectancy of greater than 12 weeks;
9. Adequate hematologic and organ function;
10. Female subjects who are not pregnant or breastfeeding
11. Male and female subjects able to have children must agree to use highly effective method of contraception throughout the study and for at least 120 days after last dose.

Exclusion Criteria:

1. Known hypersensitivity to any monoclonal antibody, QL1604 and/or any of its excipients;
2. Subjects with known central nervous system (CNS) metastasis;
3. Active autoimmune disease that has required systemic treatment in past 2 years, replacement therapy is acceptable;
4. Subjects with major cardiovascular and cerebrovascular diseases;
5. Subjects with uncontrollable pleural effusion, pericardial effusion or ascites;
6. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug;
7. Subjects who have received surgery, radiotherapy, chemotherapy, targeted therapy, other anti-tumor treatments, or participating in other clinical studies is less than 4 weeks before the first administration of investigational product;
8. Subjects who have not recovered to CTC AE Grade 1 or better from related side effects of any prior antineoplastic therapy;
9. Received a live vaccine within 30 days of planned start of study medication;
10. Infection with human immunodeficiency virus (HIV), HAV, HBV and HCV;
11. Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-ligand 1 (anti-PD-L1), anti-PD-L2 agent, cytotoxic lymphocyte associated protein-4 (CTLA-4), OX-40, CD137;
12. Known psychiatric or substance abuse disorders that would interfere with the requirements of the study;
13. History or current evidence of any condition, therapy, or laboratory abnormality, that might confound the results of the trial, or interfere with the participant's participation for the full duration of the study, or investigators/sponsor consider the subjects are not suitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate (assessed by independent radiological review committee (IRRC) per RECIST Version 1.1 and iRECIST)

SECONDARY OUTCOMES:
ORR | up to 2 years
  Objective response rate (assessed by the investigators per RECIST Version 1.1 and iRECIST)
6-month PFS rate | the proportion of subjects who have time interval over 6 months between the first dose and disease progression or death
  6-month progression-free survival (PFS) rate
6-month OS rate | from the date of first dose until the date of 6-month
  6-month overall survival rate
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier), assessed up to 2 years
  Progression-free survival (assessed by independent radiological review committee (IRRC) per RECIST v1.1 and iRECIS)
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier), assessed up to 2 years
  Progression-free survival (assessed by the investigators per RECIST v1.1 and iRECIST)
OS | from the date of first dose until the date of death from any cause， assessed up to 2 years
  Overall survival
DOR | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier), assessed up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Derived] Bi F, Dong J, Jin C, Niu Z, Yang W, He Y, Yu D, Sun M, Wang T, Yin X, Zhang R, Chen K, Wang K, Wang Z, Li W, Zhang Z, Zhang H, Guo Q, Wang X, Han L, Zhang X, Shen W, Zhang L, Ying J, Wu M, Hu W, Li Z, Li X, Feng W, Zhang B, Li L, Kang X, Guo W. Iparomlimab (QL1604) in patients with microsatellite instability-high (MSI-H) or mismatch repair-deficient (dMMR) unresectable or metastatic solid tumors: a pivotal, single-arm, multicenter, phase II trial. J Hematol Oncol. 2024 Nov 11;17(1):109. doi: 10.1186/s13045-024-01627-5. PMID 39529169